CLINICAL TRIAL: NCT06190379
Title: Aromatherapy for Upper Respiratory Health: A Randomized, Placebo Controlled, Triple-Blind Clinical Trial
Brief Title: Aromatherapy for Upper Respiratory Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Collaborators: Prodeco Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 22-12-500
Record Dates: First submitted 2022-12-05; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Immune System

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Essential oil blend in an inhaler stick
  Interventions: Other: Essential oil blend
- Placebo (Placebo Comparator): blank inhaler stick
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Essential oil blend — an aroma stick containing a blend of essential oils
  Arms: Intervention
Other: Placebo — an aroma stick containing an inert blend of oils
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm and quantify the effects of aromatherapy on respiratory health.

DETAILED DESCRIPTION:
Participants will inhale the scent from an aroma stick every waking hour for the entire duration of a period of respiratory symptoms or 14 days, whichever is shorter. As it is a randomized, placebo-controlled study, some participants will inhale the scent from an aroma stick containing active essential oils while other participants will inhale from an aroma stick containing no essential oils.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness and demonstrated ability to comply with all study procedures and availability for the duration of the study
* Gender expression: female
* Aged 20-65
* In good general health
* Exhibiting routine upper respiratory symptoms such as: sneezing, coughing, running nose, headache, general fatigue, or dry or sore throat, etc.
* Ability to utilize the inhaler and be willing to adhere to the regimen

Exclusion Criteria:

* Current use of bronchodilators or asthma medications
* Presence of asthma diagnosis or other severe breathing disorder
* Pregnant or trying to conceive
* Known allergic reactions to components of the inhaler, specifically plants in the following families: rutaceae, pinaceae, labiatae, and myrtaceae.
* Treatment with another investigational drug or other intervention within 30 days
* Current smoker
* COVID-19 diagnosis

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
severity of respiratory symptoms | 14 days
  Respiratory symptoms are measured using the Franklin Immune Scale, Respiratory Subdomain, which documents the presence of over 20 symptoms, then rates them by severity. Lower scores mean lesser severity.
duration of respiratory symptoms | daily up to 14 days
  Respiratory symptoms are measured daily; total number of days with symptoms will be calculated to produce a duration score

SECONDARY OUTCOMES:
sleep scores using the Franklin Health Sleep Scale | 14 days
  The Franklin Health Sleep Scale measures the quantity and quality of sleep across 6 subdomains. Scores are ranked on a likert scale, with higher scores indicating greater sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Hawkins, PhD, Principal Investigator — Nutraceuticals Research Institute
Locations (1):
- Franklin Health Research, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No